CLINICAL TRIAL: NCT04913792
Title: Clinical Outcomes With an Extended Range of Vision Intraocular Lens
Brief Title: Visual Performance of Multifocal Intraocular Lenses
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Clinical Professor, Wenzhou Medical University
Other Study IDs: APAC-20161013
Record Dates: First submitted 2017-11-06; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: IOL; Cataract
Keywords: multifocal IOL; ocular optical quality; abberation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ZXR00: The ZXR00 group included 30 patients bilaterally implanted with the Tecnis Symfony IOL (Abbott Medical Optics, Inc.)
  Interventions: Device: ZXR00

INTERVENTIONS:
Device: ZXR00 — This prospective comparative study included 60 eyes undergoing cataract surgery with implantation of an extended range of vision IOL.(Abbott Medical Optics, Inc.)

SUMMARY:
To evaluate the clinical outcomes with an extended range of vision (ERV) IOL based on achromatic diffractive technology.

DETAILED DESCRIPTION:
This was a prospective comparative study including 60 eyes undergoing cataract surgery with implantation of the ERV Tecnis Symfony IOL (Abbott Medical Optics, Inc.) (ERV group: 60 eyes of 30 patients). Visual, refractive, contrast sensitivity, defocus curve, ocular optical quality (Optical Quality Analysis System; iTrace), and visual function questionair（NEI-VFQ 25） outcomes were evaluated during a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* visually significant cataract
* age of 20 years or older
* preoperative corneal astigmatism of 1.50 diopters (D) or lower.

Exclusion Criteria:

* previous ocular surgery
* active ocular pathology
* amblyopia
* systemic or ocular medication that could affect vision
* subclinical or clinical corneal ectatic disease
* pupil abnormalities
* intraoperative complication leading to capsular or zonular abnormalities

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were visually significant cataract and were informed about their inclusion in the study and provided written consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-07-07 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Uncorrected distance VA（5m，66cm，40cm） | After operation （Month 3）
  logarithmic visual acuity chart

SECONDARY OUTCOMES:
Questionnaire concerning halo and visual function | After operation （Month 3）
  NEI-VFQ 25 patient questionnaire score. The questionnaire consisted of 3 parts. The first part assessed patients' satisfaction with their overall vision during the day, or at night. The score ranged from 1 to 5 (1 = not at all; 2 = a little bit; 3 = moderately; 4 = quite a bit; 5 = extremely). In part 2, patients were asked to rate the extent to which they have difficulties with their overall vision during the day or at night. The score ranged from 1 to 5 (1 = none of the time; 2 = some of the time; 3 = half of the time; 4 = most of the time; 5 = all of the time). In part 3, patients were asked to rate their overall vision and their vision at near, intermediate, and distance on a scale ranging from 0 to 10 (0 = worst; 10 = best).
abberation and kappa angle | After operation （Month 3）
  iTrace visual function analyzer
MTF cut-of and OSI | After operation （Month 3）
  MTF cut-of and OSI values measured by optical quality analysis system [OQAS]

CONTACTS AND LOCATIONS:
Overall Officials: yune zhao, MD, Study Chair — Wenzhou Medical University
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang, China

REFERENCES:
- [Result] Millan MS, Vega F. Extended depth of focus intraocular lens: Chromatic performance. Biomed Opt Express. 2017 Aug 31;8(9):4294-4309. doi: 10.1364/BOE.8.004294. eCollection 2017 Sep 1. PMID 28966865
- [Result] Kaymak H, Hohn F, Breyer DR, Hagen P, Klabe K, Gerl RH, Mueller M, Auffarth GU, Gerl M, Kretz FT. [Functional Results 3 Months after Implantation of an "Extended Range of Vision" Intraocular Lens]. Klin Monbl Augenheilkd. 2016 Aug;233(8):923-7. doi: 10.1055/s-0042-104064. Epub 2016 Jul 6. German. PMID 27385257
- [Result] Esteve-Taboada JJ, Dominguez-Vicent A, Del Aguila-Carrasco AJ, Ferrer-Blasco T, Montes-Mico R. Effect of Large Apertures on the Optical Quality of Three Multifocal Lenses. J Refract Surg. 2015 Oct;31(10):666-76. doi: 10.3928/1081597X-20150928-01. PMID 26469074
- [Result] Attia MSA, Auffarth GU, Kretz FTA, Tandogan T, Rabsilber TM, Holzer MP, Khoramnia R. Clinical Evaluation of an Extended Depth of Focus Intraocular Lens With the Salzburg Reading Desk. J Refract Surg. 2017 Oct 1;33(10):664-669. doi: 10.3928/1081597X-20170621-08. PMID 28991333
- [Result] Attia MS, Khoramnia R, Auffarth GU, Kirchner M, Holzer MP. Near and intermediate visual and reading performance of patients with a multifocal apodized diffractive intraocular lens using an electronic reading desk. J Cataract Refract Surg. 2016 Apr;42(4):582-90. doi: 10.1016/j.jcrs.2015.11.047. PMID 27113882
- [Result] Attia MS, Auffarth GU, Khoramnia R, Linz K, Kretz FT. Near and intermediate reading performance of a diffractive trifocal intraocular lens using a reading desk. J Cataract Refract Surg. 2015 Dec;41(12):2707-14. doi: 10.1016/j.jcrs.2015.06.038. PMID 26796451